CLINICAL TRIAL: NCT04327791
Title: COmbination Therapy With Baloxavir and Oseltamivir 1 for Hospitalized Patients With Influenza (The COMBO Trial 1)
Acronym: COMBO 1
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bassett Healthcare (Other)
Collaborators: Genentech, Inc. (Industry); Viroclinics Biosciences B.V. (Industry)
Responsible Party: Principal Investigator, Daniel Freilich, MD, attending physician - hospitalist, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1579493
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- baloxavir (Experimental): Baloxavir: 40 mg po once for wt < 80 kg OR 80 mg po once for wt >/= 80 kg
  Interventions: Drug: Baloxavir
- placebo (Placebo Comparator): placebo po once
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Baloxavir — administered PO once
  Arms: baloxavir
Drug: Placebos — administered PO once
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase 2-like, investigator-directed trial of hospitalized patients with laboratory confirmed influenza. Eligible and consented patients will be randomly assigned, in a 1:1 ratio, to one of two groups: Group 1, the combination treatment group (oseltamivir and baloxavir); Group 2, the standard treatment group (oseltamivir and placebo).

DETAILED DESCRIPTION:
Up to 60 hospitalized patients with laboratory confirmed influenza who provide informed consent and meet trial inclusion/exclusion criteria.

Experimental Design and Methods In a randomized, double-blind, placebo-controlled Phase 2-like, investigator-directed trial, hospitalized patients with laboratory confirmed influenza meeting inclusion and exclusion criteria, will be provided information on the trial, offered enrollment, and enrolled randomly in a 1:1 ratio to one of two groups upon signing of the study's informed consent form: Group 1, the combination treatment group (oseltamivir and baloxavir); Group 2, the standard treatment group (oseltamivir and placebo).

* Group 1, the combination treatment group will receive oseltamivir and baloxavir

  * Oseltamivir: 75 mg po bid for 5 days
  * Baloxavir: 40 mg po once for wt < 80 kg OR 80 mg po once for wt >/= 80 kg
* Group 2, the standard treatment group will receive oseltamivir and placebo

  * Oseltamivir: 75 mg po bid for 5 days
  * Placebo: Once

Oseltamivir dosing may be reduced for patients with decreased renal function as follows, per treating physician:

* CrCl > 60 mL/minute: No dosage adjustment
* CrCl > 30 to 60 mL/minute: 30 mg po bid
* CrCl > 10 to 30 mL/minute: 30 mg po qd
* HD: 30 mg po once and 30 mg po after each HD session
* CAPD: 30 mg po once
* CRRT: 30 mg po qd After assignment of a unique study number after signing informed consent, baseline data will be collected at time 0 including personal and clinical information and protocol directed laboratory specimens - nasal swabs for influenza PCR for patients who only had a rapid antigen test and blood specimens for patients who consent to additional blood drawing (for improved efficacy and safety analyses; not required for enrollment). Patients will be given oseltamivir by their healthcare providers. Research personnel's only involvement for oseltamivir dosing will be to remind providers that earlier treatment improves efficacy. Patients will then be given a single dose of baloxavir or placebo by the study's CRC as per a computerized random allocation scheme with dose determined by weight (as above); the CRC will notify the patient's provider that the patient has been given the single (blinded) dose. At time 1, 2, 3, 4, 7, and 30 days, nasal swabs will again be obtained, clinical information will be obtained from the patient via interview and review of the EMR, and blood specimens for patients who consented to additional blood drawing. Follow up will continue for 30 days.

Efficacy and adjudicated safety data points will be assessed by a Data Monitoring Committee (DMC) quarterly and as needed throughout the trial.

ELIGIBILITY:
Inclusion Criteria

1. Adults >/= 18 years old
2. Laboratory confirmed influenza A and/or B (rapid test or PCR)
3. Able to be enrolled, randomized, and dosed with study drug within 8 hours of the decision to admit patient to hospital for treatment of influenza
4. Oseltamivir treatment ordered by clinical team AND patient is able to be enrolled:

   * Prior to the initial dose of oseltamivir OR
   * Within 60 minutes after the initial dose of oseltamivir
5. Subject or Legally Authorized Representative able to and willing to provide written informed consent
6. Able to commit to 30 days of follow up
7. Weight > 40 kg
8. SARS-CoV-2 PCR swab sent within 1 week of enrollment

Exclusion Criteria

1. ESRD not undergoing hemodialysis (HD) or peritoneal dialysis (CAPD)
2. Severe hepatic insufficiency, cirrhosis, acute or chronic liver failure
3. Nausea/vomiting, aspiration risk, or other conditions precluding the ability to use oral medications (if patient is NPO including meds, otherwise unable to swallow oral medications)
4. Influenza medication use within the prior week, other than the initial oseltamivir given during this hospitalization for this episode of influenza
5. Oseltamivir or baloxavir allergy or intolerance
6. Pregnancy (need negative pregnancy test (urine or blood) in reproductive age women)
7. Absence of dependable contraception in reproductive age women
8. Inability to obtain informed consent
9. Refusal of oseltamivir therapy by patient as baseline treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-04-03 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to Clearance of Viral Shedding | 30 days
  influenza viral titer obtained by nasal swab using qCulture

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Freilich, MD, Principal Investigator — Bassett Medical Center
Locations (3):
- United States (3):
  - Baystate Medical Center, Springfield, Massachusetts
  - Bassett Medical Center, Cooperstown, New York
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No